CLINICAL TRIAL: NCT01526616
Title: Metformin Versus Metfotmin Plus Low-dose Spironolactone in the Treatment of Overweight/Obese Patients With Polycystic Ovary Syndrome: a Randomized Study
Brief Title: Spironolactone Plus Metformin in Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Prof Antonino Belfiore, Full Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010.31
Record Dates: First submitted 2012-01-27; First posted 2012-02-06 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; metformin; spironolactone; metabolic syndrome; hyperandrogenism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome; Hyperandrogenism | interventions — Metformin; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Active Comparator): 850 mg/day twice a day
  Interventions: Drug: Metformin
- Metformin plus spironolactone (Active Comparator): Metformin 850 mg twice a day for six months plus Spironolactone 25 mg day
  Interventions: Drug: Metformin plus Spironolactone

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg twice a day for six months
  Arms: Metformin
Drug: Metformin plus Spironolactone — Metformin 850 mg twice a day for six months plus Spironolactone 25 mg day
  Arms: Metformin plus spironolactone

SUMMARY:
The investigators examined whether a combined therapy with low-dose spironolactone plus metformin is more effective than metformin alone in 52 overweight/obese Polycystic Ovary Syndrome (PCOS) patients.

DETAILED DESCRIPTION:
In the present prospective, randomized study, we evaluated the efficacy of a combined therapy with metformin and low-dose spironolactone as compared to metformin alone on the clinical and endocrine-metabolic alterations of PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese patients with PCOS

Exclusion Criteria:

* Other causes of hyperandrogenism and
* Use of drugs including:

  * oral contraceptive
  * anti-hypertensive agents
  * anti-diabetic drugs
  * agents for weight loss

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Metformin versus Metformin plus low-dose Spironolactone on metabolic parameters of Patients with Polycystic Ovary Syndrome: a randomized study | six months
  We evaluated metabolic parameters across anthropometric parameters: height, weight, waist circumference, BMI, glycemia, lipid profile, blood count, coagulation parameters, hepatic and renal function indexes, OGTT and HOMA-IR. The diagnosis of MetS was established according to the ATPIII criteria

SECONDARY OUTCOMES:
Spironolactone versus Metformin plus spironolactone in hyperandrogenism in Polycystic Ovary Syndrome | six months
  We evaluated hyperandrogenism across Hirsutism Score, measuring total testosterone, SHBG, Δ4androstenedione, DHEA-S and FAI. All patients underwent ovarian ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: A. Mazza B. Fruci A. Belfiore, Doctors, Principal Investigator — Endocrinology Unit

REFERENCES:
- [Derived] Mazza A, Fruci B, Guzzi P, D'Orrico B, Malaguarnera R, Veltri P, Fava A, Belfiore A. In PCOS patients the addition of low-dose spironolactone induces a more marked reduction of clinical and biochemical hyperandrogenism than metformin alone. Nutr Metab Cardiovasc Dis. 2014 Feb;24(2):132-9. doi: 10.1016/j.numecd.2013.04.016. Epub 2013 Jul 8. PMID 23845740